CLINICAL TRIAL: NCT06206031
Title: Use of Intraosseous Doppler Ultrasonography to Study Skeletal Physiology - Echo-Os Study: Exploratory Study Before Its Use in Space Physiology
Brief Title: Intraosseous Doppler Ultrasonography to Study Skeletal Physiology: Exploratory Study Before Use in Space Physiology
Acronym: Echo-Os
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 49RC23_0347; 2023-A02403-42 (Other: ANSM)
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteers
Keywords: Bone blood circulation; Tibial cortical blood flow; Intraosseous ultrasound; Venous occlusion; Arterial occlusion
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Intervention Model Description: This small-n pilot study in physiology aims to validate the concept and serve a basis for in-depth studies on space physiology. Two clinical centers will be involved, each providing measurements in its area of expertise, and two sub-protocols with complementary objectives will be implemented:
  * Sub-protocol 1 (16 males of 20-40 yrs with usable data): Study of cortical bone vascular reactivity and its reproducibility at medial tibia (Angers University Hospital);
  * Sub-protocol 2 (16 males of 20-70 yrs with usable data): Study of bone perfusion at distal and ultradistal tibia, and comparison of bone measurements by ultrasound to those by peripheral quantitative computed tomography (Saint-Etienne University Hospital).
  Bone ultrasonography will be performed for both sub-protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- "Intraosseous ultrasonography" (Experimental): All subjects of each sub-protocol receive identical intervention (single group assignment for each of 2 sub-protocols).
  Interventions: Device: Intraosseous ultrasonography at tibia before, during, and after a physiological vascular stimulation (venous occlusions, arterial occlusion, handgrip)

INTERVENTIONS:
Device: Intraosseous ultrasonography at tibia before, during, and after a physiological vascular stimulation (venous occlusions, arterial occlusion, handgrip) — Timing for sub-protocol 1 (performed twice with 2-to-10-day interval): donning in supine position - rest 5 minutes - venous occlusion to 40 mmHg 3 minutes - rest 10 minutes - arterial occlusion to 200mmHg 2 minutes - post-occlusion period 10 minutes - rest 10 minutes - static handgrip 30% Maximum Voluntary Force 3 minutes - recovery 2 minutes and doffing.
  Timing for sub-protocol 2 (performed once). First, two sequences of intraosseous ultrasonography are performed in 45° head-up tilt position, with 10-minutes rest between sequences: donning and rest 5 minutes - occlusion to 80 mmHg 2 minutes - rest 10 minutes - occlusion to 180 mmHg 2 minutes - rest 10 minutes. During the first sequence, ultrasonography probe is positioned between middle and lower third of tibia for cortical bone measurement; during the second - at distal epiphysis of the tibia for trabecular bone measurement. After ultrasonography, subject is sitting down for 10 minutes for computed tomography.

SUMMARY:
Use of intraosseous Doppler ultrasonography to study skeletal physiology ("Echo-Os Study"). Exploratory study before its use in space physiology.

Bones have a complex vascular network providing nutrients and oxygen to bone cells. The physiology of intraosseous blood circulation remains very little known to date, particularly in human. Human bone vascularization studying is very difficult because of a lack of simple tools for functional exploration of bone vascular perfusion. For blood flow studies, ultrasonography is best suited, allowing for dynamic non-invasive measures. Bone has until now been considered to stop ultrasound and therefore prevent any intraosseous measurements. From a physics viewpoint, bones conduct ultrasound waves well, but they are reflected differently compared to soft tissues. A specific analysis of the ultrasound returned by the bone, using specific correction factors, is therefore needed to interpret ultrasound signals, reconstruct an anatomical image, and extract physiological information. The system proposed in this study combines standard conventional low-frequency ultrasound probes with a specific analysis of ultrasound wave reflection. This system makes it possible to reconstruct an anatomical bone image and record the pulsatile signal of intraosseous vascular perfusion. The investigators will use this system to study the vascular reactivity induced by different physiological maneuvers.

This protocol proposes to study the following mechanisms of blood flow regulation at the level of tibia cortical bone: flow-mediated dilation induced by endothelium (with arterial occlusion test), vasoconstriction induced by sympathetic activation (with static handgrip test), and vasoconstriction induced by veno-arteriolar reflex (with venous occlusion test). This is a pilot study in physiology performed with healthy volunteers. This study will verify whether our intraosseous ultrasound system can properly measure physiological responses expected during these maneuvers. This protocol will also establish links between perfusion and bone architecture at tibial level.

ELIGIBILITY:
Inclusion Criteria for sub-protocol 1:

* Male aged 20-40 years

Inclusion criteria for sub-protocol 2:

* Male aged 20-40 years & 50-70 years
* Body height of at least 180 cm (in order to have tibia length of 43-45 cm allowing the positioning of ultrasonic probe at distal tibia, and occlusive cuff at calf level)
* Bone densitometry with available report performed within 5 last years (if none has been done, possibility to perform densitometry covered by the study at selection or inclusion visit)

Inclusion criteria common for both sub-protocols:

* Healthy volunteer without chronic pathology (in particular no known rhythm disorder) or long-term treatment
* No symptomatic acute medical event requiring treatment on the visit days
* No history of tibia fractures
* Body Mass Index between 19 and 26
* Affiliation to the French Social Security System
* Written informed consent

Non-Inclusion criteria:

* Inability to stay still for 20 minutes (tremor)
* Active smoking (stopped less than 1 year ago)
* History of prolonged corticosteroid treatment
* Deprivation of liberty by legal or administrative decision
* Subject to involuntary psychiatric treatment
* Subject to a legal protection measure
* For sub-study 1: Osteoporosis known at interview

Exclusion Criteria:

* Any abnormality or deviation from the selection criteria identified during the clinical examination at the inclusion visit (non-sinus rhythm in ECG, body temperature > 38°C, blood pressure or heart rate outside the defined standards, etc.)

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Change in tibial intracortical blood flow velocity, induced by physiological maneuvers in supine position (sub-protocol 1) | before, at the end of venous occlusion (40 mmHg 3 minutes); before, at the end of arterial occlusion (200 mmHg 2 min); at 2, 5, and 10 min of post-occlusion period; before, at the end of handgrip (30% maximum voluntary force for 3 minutes)
  Velocity (mm/s) of intracortical blood flow at medial tibia level and its response to venous occlusion, arterial occlusion, handgrip, will be assessed via Ultrasound Vector Flow Mapping

SECONDARY OUTCOMES:
Change in leg skin and muscle blood flow, induced by physiological maneuvers in supine position (sub-protocol 1) | before, at the end of venous occlusion (40 mmHg 3 minutes); before, at the end of arterial occlusion (200 mmHg 2 min); at 2, 5, and 10 min of post-occlusion period; before, at the end of handgrip (30% maximum voluntary force for 3 minutes)
  Leg skin blood flow (arbitrary units), leg muscle change in concentrations of oxy- and deoxy-hemoglobin (µmol/L), and their responses to venous occlusion, arterial occlusion, handgrip, will be assessed via Laser Doppler flowmetry and Near-Infrared Spectroscopy
Comparison of changes in tibial intracortical blood flow with changes in leg skin and muscle blood flow, induced by physiological maneuvers in supine position (sub-protocol 1) | before, at the end of venous occlusion (40 mmHg 3 minutes); before, at the end of arterial occlusion (200 mmHg 2 min); at 2, 5, and 10 min of post-occlusion period; before, at the end of handgrip (30% maximum voluntary force for 3 minutes)
  Responses of leg intracortical, skin, and muscle blood flow to venous occlusion, arterial occlusion, and handgrip will be expressed as % baseline. Correlation of bone responses to skin and muscle responses (Pearson r) will be calculated.
Reproducibility of the change in tibial intracortical blood flow velocity, induced by physiological maneuvers in supine position (sub-protocol 1) | before, at the end of venous occlusion (40 mmHg 3 minutes); before, at the end of arterial occlusion (200 mmHg 2 min); at 2, 5, and 10 min of post-occlusion period; before, at the end of handgrip (30% maximum voluntary force for 3 minutes)
  Measurements for sub-protocol 1 will be performed 2 times (visit 1 and visit 2 with 2-to-10-day interval), and Coefficient of variation in responses to physiological maneuvers (%) will be calculated
Change in tibial intracortical blood flow velocity, induced by occlusion maneuvers in +45° head up tilt position (sub-protocol 2) | Ultrasonography acquisition sequences of 5 secondes will be performed before and during each occlusions.
  Velocity (mm/s) of intracortical blood flow at distal tibia level, and its responses to proximal cuff compression steps of 80 mmHg and 180 mmHg, will be assessed via Ultrasound Vector Flow Mapping.
Change in tibial ultradistal bone blood flow velocity, induced by occlusion maneuvers in +45° head up tilt position (sub-protocol 2) | Ultrasonography acquisition sequences of 5 secondes will be performed before and during each occlusions.
  Velocity (mm/s) of intracortical blood flow at distal tibia level, and its responses to proximal cuff compression steps of 80 mmHg and 180 mmHg, will be assessed via Ultrasound Vector Flow Mapping.
Comparison of intraosseous ultrasonography and computed tomography for Cortical bone thickness characterisation (sub-protocol 2) | First, intraosseous ultrasonography is performed at +45° head up tilt position (30 minutes for all occlusion steps), then the subject sits down and tomography is performed (10 minutes)
  Cortical thickness at distal tibia (mm) will be measured via peripheral quantitative computed tomography and via intraosseous ultrasonography. Correlation (Pearson r) between measurements will be calculated
Comparison of intraosseous ultrasonography and computed tomography for Cortical bone porosity characterisation (sub-protocol 2) | First, intraosseous ultrasonography is performed at +45° head up tilt position (30 minutes for all occlusion steps), then the subject sits down and tomography is performed (10 minutes)
  Cortical density (mg/cm3) via peripheral quantitative computed tomography and cortical ultrasound propagation velocity (m/s) via intraosseous ultrasonography will be measured at distal tibia. Correlation (Pearson r) between measurements will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Antoine CUSTAUD, Professor, Principal Investigator — University Hospital, Angers
Locations (2):
- France (2):
  - CHU d'Angers, Angers
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).